CLINICAL TRIAL: NCT00001889
Title: Comparison of Myocardial Contrast Echo With Dobutamine Echo in Diagnosis of Coronary Artery Disease
Brief Title: Comparison of Echocardiographic Techniques in Diagnosis of Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990077; 99-H-0077
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-02

CONDITIONS: Coronary Disease
Keywords: Microbubbles; Myocardial Blood Flow; Myocardial Ischemia; Second Harmonics; Ultrasound; Coronary Artery Disease
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Coronary Artery Disease | interventions — Dobutamine

INTERVENTIONS:
Procedure: Myocardial contrast echocardiography
Procedure: Stress echocardiography with dobutamine

SUMMARY:
This study is designed to compare two different echocardiographic techniques in the evaluation of heart disease (coronary artery disease). Both tests called Myocardial Contrast Echocardiography with Pharmacologic Stress and Stress Echocardiography with Dobutamine, are performed using a standard echocardiographic machine.

Myocardial Contrast Echocardiography (MCE) does not use radioactivity. It uses sound waves like standard echocardiography. However, with MCE patients receive an injection of a "contrast agent" directly into the blood stream through a vein. The contrast agent, called Optison, is made of tiny microbubbles smaller than red blood cells. The echocardiogram can detect these microbubbles in the small blood vessels of the heart muscle and allow researchers to find areas of the heart receiving less blood flow than others. It is important to observe the heart during exercise because there are changes in blood flow. Since MCE cannot be performed when the patient is exercising, researchers give medication (adenosine) that stimulates the heart and creates a situation similar to exercise.

Stress Echocardiography with Dobutamine does not use radioactivity. It uses sound waves like standard echocardiography. During this echocardiogram patients receive doses of a medication called dobutamine that stimulates the heart to beat stronger and faster.

The purpose of this study is to evaluate the accuracy of MCE compared to stress echocardiography at detecting coronary artery disease (CAD).

DETAILED DESCRIPTION:
Stress echocardiography has become a valuable technique for the non-invasive detection of coronary artery disease (CAD). Its accuracy has been shown to be superior to that of the exercise electrocardiogram and comparable to that of myocardial perfusion imaging. Myocardial contrast echocardiography (MCE) offers the potential to evaluate tissue perfusion at the level where oxygen transfer to the myocytes occurs. MCE can, therefore, provide information regarding the functional status of the myocardial microvasculature and presence of blood flow disparity. The purpose of this study is to evaluate the accuracy of MCE compared to stress echocardiography. We will correlate these results with findings from coronary angiography and compare the ability of those techniques to detect CAD.

ELIGIBILITY:
Patients with known or suspected coronary artery disease.

Adults 18 years of age or older.

No pre-menopausal patients who are lactating, pregnant or potentially pregnant as judged by history, physical examination, ultrasound or urine pregnancy test.

No unstable angina patients.

No recent myocardial infarction patients (less than 1 month).

No frequent ectopy which precludes adequate image acquisition.

No history of asthma or chronic obstructive pulmonary disease.

No patients receiving aminophylline, theophylline or dipyridamole.

No presence of second and third degree heart block without pacemaker.

No significant hypertension (systolic blood pressure greater than 170 mm Hg) or hypotension (systolic blood pressure less than 100 mm Hg).

No hypotension: basal sitting systolic arterial pressure less than 100 mm Hg confirmed 30 minutes later.

No sinus tachycardia greater than or equal to 100 beats per min.

No atrial fibrillation.

No inadequate two-dimensional echocardiographic windows.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1999-03; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lumley P, Broadley KJ, Levy GP. Analysis of the inotropic: chronotropic selectivity of dobutamine and dopamine in anaethetised dogs and guinea-pig isolated atria. Cardiovasc Res. 1977 Jan;11(1):17-25. doi: 10.1093/cvr/11.1.17. PMID 12867
- [Background] Armstrong WF. Stress echocardiography for detection of coronary artery disease. Circulation. 1991 Sep;84(3 Suppl):I43-9. PMID 1884503
- [Background] Pellikka PA. Stress echocardiography in the evaluation of chest pain and accuracy in the diagnosis of coronary artery disease. Prog Cardiovasc Dis. 1997 May-Jun;39(6):523-32. doi: 10.1016/s0033-0620(97)80011-4. PMID 9166363